CLINICAL TRIAL: NCT06401993
Title: Peripheral-central Correlation Study on the Treatment of Chronic Tinnitus With "Dao qi Tong Luo" Based on the Theory of "Connecting the Two Ears to the Brain"
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jie Zhou, Principal Investigator, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSLL-KY-2024-038-01
Record Dates: First submitted 2024-04-30; First posted 2024-05-07 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Tinnitus
Keywords: Acupuncture; Fnirs; Tinnitus; ABR
MeSH Terms: conditions — Tinnitus

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The "dao qi tong luo" group (Experimental): Subjects in the "dao qi tong luo" group will undergo acupuncture treatment, which is administered 10 times
  Interventions: Procedure: The "dao qi tong luo" group
- The acupuncture group (Sham Comparator): Subjects in the acupuncture group will undergo acupuncture treatment, which is administered 10 times
  Interventions: Procedure: The acupuncture group

INTERVENTIONS:
Procedure: The "dao qi tong luo" group — The "dao qi tong luo" group will accept acpuncture. Acupuncture will be performed at acupoints including TE17 (Yifeng), SI19 (Tinggong), GB2 (Tinghui), TE5 (Waiguan), TE3 (Zhongzhu) and etc. Among them, the "dao qi tong luo" group will make patients feel qi.
  Arms: The "dao qi tong luo" group
Procedure: The acupuncture group — The acupuncture group will accept acpuncture. Acupuncture will be performed at acupoints including TE17 (Yifeng), SI19 (Tinggong), GB2 (Tinghui), TE5 (Waiguan), TE3 (Zhongzhu) and etc. The acupuncture group will not feel qi.
  Arms: The acupuncture group

SUMMARY:
By comparing the clinical manifestations, ABR parameters and cerebral cortex blood oxygen levels of chronic tinnitus patients and healthy subjects under two different body states, the peripheral-central correlation of chronic tinnitus patients was explored, and the modern scientific significance of the theory of "two ears connecting the brain" was initially expounded. On this basis, the immediate and cumulative effects and peripheral-central correlation of "dao qi tong luo" intervention in chronic tinnitus were observed, and the effective mechanism of "dao qi tong luo" treatment was explored.

DETAILED DESCRIPTION:
The study will enroll 15 healthy subjects and 72 subjects with chronic tinnitus. Functional near infrared spectroscopy (fNIRS) will be used to examine specific brain regions, and ABR techniques will record auditory brainstem responses in chronic tinnitus patients and healthy subjects. Lateral comparison was made between chronic tinnitus patients and healthy subjects on the parameters of auditory brainstem response and the level of oxygen outside the cerebral cortex, and the data of the two were integrated to conduct correlation analysis and correlation analysis with clinical manifestations, so as to compare the correlation between peripheral and central auditory function in different body states. Subsequently, the chronic tinnitus subjects will undergo a course of acupuncture treatment. At the end of acupuncture and moxibustion treatment, the immediate and cumulative effects and peripheral - central correlation of "dao qi tong luo" intervention in chronic tinnitus were observed, and the effective mechanism of "dao qi tong luo" treatment was explored.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria for patients with chronic tinnitus

  1. Chronic tinnitus patients, that is, the course of disease ≥6 months;
  2. No contraindications of fNIRS scanning;
  3. The age of 20 years ≤55 years old, gender is not limited, right-handed;
  4. The external ear canal is unobstructed and the eardrum is intact
  5. The average hearing threshold of both ears is <35dB;
  6. Normal expression and understanding ability. Inclusion criteria for healthy subjects

  <!-- -->

  1. No tinnitus, no hearing disorders and other ear diseases;
  2. Good health condition, no history of mental disease and nervous system disease;
  3. No contraindications of fNIRS scanning;
  4. The age of 20 years ≤55 years old, gender is not limited, right-handed;
  5. The external ear canal is unobstructed, and the tympanic membrane is complete;
  6. Normal expression and understanding ability.

Exclusion Criteria:

* 1.A history of drug dependence or alcohol addiction; 2.Serious central system diseases or other systemic diseases such as cardiovascular and cerebrovascular diseases; 3. Patients with organic diseases such as craniocerebral trauma; 4. Sudden deafness, Meniere's disease, otosclerosis, acoustic neuroma and other inner ear or auditory nerve diseases; 5.External otitis, acute/chronic otitis media and other external ear middle-ear related diseases; 6. Patients with auditory hypersensitivity; 7. Pregnancy, preparation for pregnancy, breastfeeding population; 8. There are metal implants in the body, fNIRS detection contraindicated.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-05-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Tinnitus Handicap Inventory (THI) | at baseline (pre-treatment),procedure
  Tinnitus Handicap Inventory is based on relevant expert consensus. THI scores range from 0 to 100, with the higher the score, the more severe the condition

SECONDARY OUTCOMES:
Tinnitus Evaluation Questionnaire (TEQ) | at baseline (pre-treatment), procedure
  Tinnitus Evaluation Questionnaire is based on relevant expert consensus. TEQ scores range from 0 to 21, with the higher the score, the more severe the condition
Auditory Brainstem Response (ABR) | at baseline (pre-treatment), procedure
  Auditory Brainstem Response is based on relevant expert consensus
Functional Near-Infrared Spectroscopy (Fnirs) | at baseline (pre-treatment), procedure
  Functional Near-Infrared Spectroscopy is based on relevant expert consensus

CONTACTS AND LOCATIONS:
Overall Officials: Jie Zhou, M.D, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jiang D, Huang XH, Fang K, Zhao MH, Li Y, Hu HT, Fang LQ, Gao H, Zhou J. Peripheral-central correlation study of acupuncture for chronic tinnitus study protocol for a randomized controlled trial. Front Med (Lausanne). 2025 Feb 13;12:1543023. doi: 10.3389/fmed.2025.1543023. eCollection 2025. PMID 40018352